CLINICAL TRIAL: NCT00875056
Title: A Phase II Study of MK-0683 in Patients With Relapsed / Refractory Follicular Lymphoma (FL), Other Indolent B-cell Non-Hodgkin's Lymphoma (B-NHL) or Mantle Cell Lymphoma (MCL)
Brief Title: Study of Vorinostat (MK-0683) With Follicular Lymphoma (FL), Other Indolent B-cell Non-Hodgkin's Lymphoma (B-NHL), or Mantle Cell Lymphoma (MCL) Participants (MK-0683-103)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-103; 2009_570; 132248 (Registry Identifier: JAPIC-CTI); MK-0683-103 (Other: Merck Protocol Number)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Vorinostat

STUDY DESIGN:
Intervention Model Description: All participants received the same drug regimen but were allocated to groups based on disease type.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Follicular Lymphoma (FL) (Experimental): Participants with relapsed/refractory FL received 200 mg of vorinostat (MK-0683) twice daily (200 mg x 2/day) for 14 consecutive days followed by 1 week (7 days) rest in a 21-day cycle, until they met the per-participant discontinuation criteria specified by the protocol.
  Interventions: Drug: Vorinostat
- Indolent non-FL B-NHL or MCL (Experimental): Participants with indolent non-follicular lymphoma (FL) B-cell non-Hodgkin's lymphoma (B-NHL), or with mantle cell Lymphoma (MCL) received 200 mg of vorinostat (MK-0683) twice daily (200 mg x 2/day) for 14 consecutive days followed by 1 week (7 days) rest in a 21-day cycle, until they met the per-participant discontinuation criteria specified by the protocol.
  Interventions: Drug: Vorinostat
- Other Disease (Experimental): Participants with disease other than relapsed/refractory follicular lymphoma (FL), non-FL B-cell non-Hodgkin's lymphoma (B-NHL), or mantle cell Lymphoma (MCL), as assessed by the Independent Central Pathological Committee, received 200 mg of vorinostat (MK-0683) twice daily (200 mg x 2/day) for 14 consecutive days followed by 1 week (7 days) rest in a 21-day cycle, until they met the per-participant discontinuation criteria specified by the protocol. This group was created to include participants who enrolled, but whose later diagnoses by the Independent Central Pathological Committee excluded them from analysis in the FL and non-FL B-NHL/MCL groups because they had different disease than those prespecified in the protocol.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Two 100 mg oral capsules of vorinostat, twice daily (400 mg/day), on Days 1 through 14 of each 21 day cycle
  Other Names: MK-0683; Zolinza

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of vorinostat (MK-0683) in participants with relapsed and/or refractory follicular lymphoma. The exploratory purpose of this study is to evaluate efficacy of MK-0683 in participants with relapsed/refractory non-FL indolent B-NHL or relapsed/refractory MCL. The primary hypothesis is that MK-0683 will show efficacy in relapsed/refractory FL patients as measured by the Overall Response Rate.

ELIGIBILITY:
Inclusion Criteria:

* Participant has an histopathologically confirmed follicular lymphoma (FL), or other indolent B-cell non-Hodgkin's lymphoma (B-NHL) or mantle cell lymphoma (MCL)

  * Only relapsed/refractory FL can be included outside Japan
* Participant has at least one measurable lesion by computerized tomography (CT) scan which is defined by Cheson's 1999 criteria
* Participant has received at least 1 but up to 4 prior chemotherapeutic regimens, the most recent therapy must have failed to induce a partial response, or there must be recurrence in case of the most recent therapy has shown complete response, or there must be relapse in case of the most recent therapy has shown partial response
* Life expectancy of >4 months
* Participant must have adequate organ and marrow function
* Women of child bearing potential must be negative for pregnancy and agree to use effective contraceptive measures until 30 days after the last dose of MK-0683.
* Men must agree to use effective contraceptive measures until 6 months after the last dose of MK-0683

Exclusion Criteria:

* Participant has undergone allogenic transplant treatment or autologous stem cell transplant within 6 months
* Participant with other active malignancies or central neurological infiltration with lymphoma
* Participant with severe hepatic insufficiency
* Participant with history of allergic reactions attributed to any component of MK-0683
* Participant is known to be human immunodeficiency virus (HIV) antibody-, hepatitis B virus antigen- or hepatitis C virus antibody-positive
* Participant has undergone prior/concomitant treatment with MK-0683 or other histone deacetylase (HDAC) inhibitors

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2011-09-06 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ogura M, Ando K, Suzuki T, Ishizawa K, Oh SY, Itoh K, Yamamoto K, Au WY, Tien HF, Matsuno Y, Terauchi T, Yamamoto K, Mori M, Tanaka Y, Shimamoto T, Tobinai K, Kim WS. A multicentre phase II study of vorinostat in patients with relapsed or refractory indolent B-cell non-Hodgkin lymphoma and mantle cell lymphoma. Br J Haematol. 2014 Jun;165(6):768-76. doi: 10.1111/bjh.12819. Epub 2014 Mar 12. PMID 24617454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
Started | 39 | 11 | 6
Completed | 5 | 2 | 0
Not Completed | 34 | 9 | 6
Not completed — Adverse Event | 8 | 1 | 2
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Progressive Disease | 20 | 8 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease | Total
Number analyzed (Participants) | 39 | 11 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (10.4) | 62.9 (9.7) | 56.3 (10.5) | 58.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 4 | 2 | 30
  Male | 15 | 7 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 11 | 6 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 39 | 11 | 6 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Normal liver/spleen physical exam, all lymph nodes and nodal masses are normal, and there is no bone marrow involvement), a Complete Response/unconfirmed (CRu: Normal liver/spleen physical exam, plus at least a 75% decrease in the sum of the products of the greatest diameters of nodal masses if any are greater than 1.5 cm in their greatest diameter, normal or indeterminate bone marrow involvement), or a Partial Response (PR: Either normal physical exam, lymph nodes, and lymph node masses plus positive bone marrow involvement; OR normal physical exam or decrease in liver/spleen size plus at least a 50% decrease in the diameters of lymph nodes and nodal masses) as assessed using the international working group Non-Hodgkin's lymphoma standardized response criteria described by Cheson, BD in 1999. The percentage of participants who experienced a CR, CRu, or PR is presented.
Time Frame: Up to 650 days
Population: The analysis population included all allocated participants with follicular lymphoma (FL), non-FL B cell non-Hodgkin's lymphoma (B-NHL), or mantle cell lymphoma (MCL) who received at least one dose of study drug, and had some post-allocation endpoint data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
Number analyzed (Participants) | 39 | 11 | 0
Percentage of participants | 48.7 [32.4 to 65.2] | 27.3 [6.0 to 61.0] |

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE was presented.
Time Frame: Up to approximately 29 months
Population: All allocated participants who received a dose of study drug were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
Number analyzed (Participants) | 39 | 11 | 6
Participants | 39 | 11 | 6

3. Secondary Outcome: Time to Treatment Failure for Relapsed/Refractory FL
Description: Time to Treatment Failure is defined as the time from allocation until the date of any treatment failure, including documented disease progression, or discontinuation of the study medication for any reason. Data was censored on the efficacy data cutoff date of 25 February, 2011.
Time Frame: Up to 650 days
Population: The analysis population included all allocated participants with FL who received at least one dose of study drug, and had some post-allocation endpoint data.
Measure: Median (Full Range); unit: Days
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
Number analyzed (Participants) | 39 | 0 | 0
Days | 323 [60 to NA] — For time to treatment failure upper limit, not all participants had experienced a response by the time of efficacy data cutoff, making the data not available. |  |

4. Secondary Outcome: Time to Response for Relapsed/Refractory FL
Description: Time to Response is defined as the time from allocation until the time of an initial response. Data was censored on the efficacy data cutoff date of 25 February, 2011.
Time Frame: Up to 650 days
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
Number analyzed (Participants) | 39 | 0 | 0
Days | NA [NA to NA] — Median time to response not reached. For upper and lower limits, not all participants had experienced a response by the time of efficacy data cutoff, making the data not available. |  |

5. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to Experiencing an Adverse Event (AE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued from study drug due to an adverse event was reported.
Time Frame: Up to 536 days
Population: All allocated participants who received a dose of study drug were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
Number analyzed (Participants) | 39 | 11 | 6
Participants | 6 | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to approximately 65 months
Description: Non-serious adverse events and serious adverse events were counted starting at the time of a participant's first treatment and included all treated participants. All-Cause Mortality was counted starting from the time of a participant's enrollment and included all randomized participants.
Arm/Group | Follicular Lymphoma (FL) | Indolent Non-FL B-NHL or MCL | Other Disease
All-Cause Mortality (participants affected / at risk) | 9/39 | 4/11 | 3/6
Serious Adverse Events (participants affected / at risk) | 15/39 | 4/11 | 2/6
Other Adverse Events (participants affected / at risk) | 39/39 | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follicular Lymphoma (FL) (N=39) | Indolent Non-FL B-NHL or MCL (N=11) | Other Disease (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follicular Lymphoma (FL) (N=39) | Indolent Non-FL B-NHL or MCL (N=11) | Other Disease (N=6)
Anaemia (Blood and lymphatic system disorders) | 12 (25) | 5 (11) | 1 (1)
Erythropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 20 (107) | 8 (45) | 3 (11)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 13 (40) | 7 (20) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 29 (177) | 7 (89) | 2 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 37 (194) | 10 (79) | 5 (15)
Palpitations (Cardiac disorders) | 5 (6) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (9) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (8) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 3 (7) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (33) | 4 (11) | 1 (1)
Dental caries (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 28 (331) | 9 (131) | 5 (15)
Dry mouth (Gastrointestinal disorders) | 4 (10) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (6) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (8) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (97) | 7 (12) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 9 (29) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (50) | 1 (1) | 2 (4)
Asthenia (General disorders) | 6 (18) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (7) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (4) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 22 (104) | 5 (14) | 2 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 3 (3) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 (34) | 3 (10) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (60) | 4 (15) | 1 (1)
Oral herpes (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (33) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 9 (9) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 11 (27) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 12 (27) | 4 (7) | 1 (2)
Blood bilirubin increased (Investigations) | 3 (9) | 2 (4) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 10 (42) | 2 (7) | 2 (7)
Blood lactate dehydrogenase increased (Investigations) | 5 (9) | 2 (15) | 2 (7)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 4 (9) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 11 (12) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 27 (141) | 6 (15) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (15) | 0 (0) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 7 (22) | 3 (20) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (21) | 4 (7) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (13) | 3 (14) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 5 (22) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (25) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (16) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (12) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (34) | 1 (10) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (7) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (7) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (66) | 3 (5) | 3 (3)
Headache (Nervous system disorders) | 7 (12) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (4) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (2)
Proteinuria (Renal and urinary disorders) | 6 (13) | 2 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 (16) | 1 (4) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (19) | 4 (4) | 2 (2)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 9 (13) | 2 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (5) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.